## Reducing Overuse of Antibiotics at Discharge Home (ROAD Home)

NCT06106204

Consent Document for Interviews with hospital champions and stakeholders:

Consent\_Interview\_Champion\_Stakeholder\_6.22.23 V1. 06.22.2023

## **Consent Cover Letter**

The purpose of the study is to understand hospital's experience implementing the ROAD Home Intervention to reduce antibiotic overuse at hospital discharge. The ROAD Home Intervention is an antibiotic stewardship quality improvement strategy designed to support hospitals in selecting and implementing evidence-based stewardship strategies tailored to their resources and goals. We hope this research will be useful in identifying factors that facilitate the implementation of antibiotic stewardship interventions which will ultimately improve patient care.

If you agree, you will participate in a virtual (via Zoom) semi-structured interview. The purpose of the interview is to identify barriers and facilitators to implementation and to assess acceptability, feasibility, and sustainability of the ROAD Home Intervention. Interviews will be conducted by Dr. Julia E. Szymczak using a guide with additional questions tailored to your hospital based on information gathered during the intervention period.

We expect this interview to take about 1 hour. Your participation is completely voluntary. You may choose not to answer a question and are free to withdraw consent and discontinue participation in the interview at any time for any reason without penalty or loss of benefits.

The risks of participating in this interview are minimal. We will not ask you about sensitive topics, but it is possible that you may feel uncomfortable answering some questions; you may choose not to answer. There is a small risk of loss of confidentiality. This interview will be recorded and transcribed, but your name and other identifying details will not be part of these records. All data for this project will be stored on secure computer systems. You will not be identified in any publications.

If you complete this interview, you will receive a \$100 gift card for your time.

If you have any questions, complaints, or if you feel you have been harmed by this project, you may contact Dr. Valerie Vaughn, Division of General Internal Medicine at: <a href="mailto:Valerie.vaughn@hsc.utah.edu">Valerie.vaughn@hsc.utah.edu</a>.

Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at irb@hsc.utah.edu.

Research Participant Advocate: You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at participant.advocate@hsc.utah.edu.

By participating in the interview, you are giving your consent to participate in this research and to be audio-recorded. Thank you for your willingness to participate!



University of Utah Institutional Review Board Exemption 7/7/2023